CLINICAL TRIAL: NCT04578704
Title: Stability of Bimaxillary Proclination Cases Following Fixed Appliances Treatment: A Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Norhidayah Mohd Tahir, Dr.Norhidayah bt Mohd Tahir, Lecturer, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bimaxillary Proclination
Record Dates: First submitted 2020-09-25; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Bimaxillary Proclination
Keywords: stability; retainers

STUDY DESIGN:
Intervention Model Description: This study will be encompassed 3 groups of patients that will be assigned for 3 types of retention methods;
  1. VFR (upper and lower arches)
  2. Fixed bonded retainers (upper and lower arches)
  3. Double regime (bonded retainers & VFR for upper and lower arches). (Abd Rahman 2016)
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be decided for the type of retention treatment by picking an opaque and sealed envelope.
  The participants study models will be examined and assigned with a blinding code by first researcher , who will be blinded to the subjects' retainer allocation. Patients name on the printed radiograph will also be removed. Therefore,the first researcher will be blinded to those she will be measuring. The blinding code will be prepared by second researcher before first researcher measure the casts and radiographs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vacuum formed retainer group (Experimental): It will be constructed following manufacturer's instructions for the thickness.
  Interventions: Other: Vacuum formed retainer, fixed bonded retainer, vacuum formed and fixed bonded retainer
- Fixed bonded retainer group (Experimental): fixed bonded wire will be bonded on individual tooth extended distal to extraction space that were previously closed by fixed appliances treatment.
  Interventions: Other: Vacuum formed retainer, fixed bonded retainer, vacuum formed and fixed bonded retainer
- Vacuum formed retainer and fixed bonded retainer (Experimental): Double regime retainer that will be consisted of bonded retainer and vacuum formed retainer for upper and lower arch.
  Interventions: Other: Vacuum formed retainer, fixed bonded retainer, vacuum formed and fixed bonded retainer

INTERVENTIONS:
Other: Vacuum formed retainer, fixed bonded retainer, vacuum formed and fixed bonded retainer — Patients will be instructed to wear the removable vacuum form retainer for 8 to 10 hours per day and only removed the retainers during tooth brushing. (Thickett 2010), (Gill 2007).
  The vacuum formed retainer will be constructed using thermoplastic material that will be purchased from manufacturer at 1.0mm thickness.
  Meanwhile, bonded retainer will be done using Ormco ® response deadsoft retainer wire size 0.190 round, made in USA by ORMCO Corporation, the fixed bonded wire will be extended distal to the extraction spaces that were previously closed by fixed appliances on both the upper and lower arches. The bonded retainer will be wearing by patients for 24 hours.
  Double regime retainer that will be comprised of vacuum formed and bonded retainer will be constructed using the same properties as vacuum formed retainer and bonded retainer. A standard oral and written instruction will be given to patients regarding retainer's uses. (Shawesh M et.al, 2009).

SUMMARY:
Bimaxillary dental proclination is the condition where the upper and lower dental arches are procline thus increase lip fullness. Since the aim of orthodontic treatment in bimaxillary proclination in to get flatten profile where the incisor inclinations are purposely reduced or interincisal angle are increased, therefore it is guarded for corrected dentition to maintain stable or not post orthodontic treatment.Therefore, this study is looking into evidence which is the best retainer to maintain stability of bimaxillary proclination cases following fixed appliances treatment.

DETAILED DESCRIPTION:
Study title Stability of Bimaxillary Proclination Cases Following Fixed Appliances Treatment: A Randomized Control Trial

Study Population Pre-treatment of bimaxillary proclination patient who completed active orthodontic treatment with fixed appliances and are scheduled to debond at Orthodontic Clinic, Faculty of Dentistry, University of Malaya.

Study Design Randomized, prospective, single-center control trial. Three parallel arm groups of patients will be assigned for 3 types of retention methods; 1.VFR 2.Fixed bonded retainer 3.Double regime (bonded & VFR)

Aim of study To determine the best mode of retention to maintain the stability of bimaxillary proclination cases treated by four premolars extraction and fixed appliances.

Specific Objectives

1. To measure the post treatment dental and soft tissue stability in the retention phase up to one-year post treatment
2. To compare the effectiveness the different types of retainers to maintain the stability of orthodontically corrected bimaxillary proclination
3. To determine the impact of the different types of retainers on the OHRQoL

Sample Size The sample size calculation was done using G*power software version 3.1.The f-test, repeated measures ANOVA, within-between interaction were used.

Based on the effect size of 0.43 (Keating PJ 1986), maximum accuracy (power) of 80% (0.80), error of 5% (0.05), number of groups are 3, number of measurements are 2, correlation among repetitive measures is 0.5, nonsphericity correlation is 1, total number of 18 subjects needed for entire study. Allowing for 50% dropout, a final sample size of 27 subjects with 9 subjects per group will be used.

Study Duration September 2019 - Disember 2021

ELIGIBILITY:
Inclusion Criteria:

1. Pretreatment bimaxillary proclination patients with interincisal angle less than 125º (Keating PJ 1986).
2. Patients with fixed orthodontic appliances treatment on both arches consisting of the extraction of 4 premolars (Keating 1986).
3. Both arches are indicated for retainers.
4. Pre-treatment lateral cephalometric radiograph of adequate diagnostic quality.

Exclusion Criteria:

1. Pretreatment spacing eg: Median diastema.
2. No change or proclined lower labial segment post treatment.
3. Early debond patient.
4. Patient intended to relocate within study period.
5. Hypodontia that require prosthesis, cleft lip and/or cleft palate, or orthognathic cases.
6. Patients with learning disabilities and unable to listen, speak and read written instructions in Bahasa Melayu or English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Stability: Change in the incisal inclinations | 1 year post debond of orthodontic fixed appliances
  To measure any changes in the upper incisor to maxillary plane angle, lower incisor to mandibular plane angle and changes in interincisal angle. This angular measurement will be measured in degree.

SECONDARY OUTCOMES:
Stability: Soft tissue changes | 1 year post debond of orthodontic fixed appliances
  To measure any changes in the nasolabial angle, labiomental angle. These will be measured in degree. The upper and lower lips distances in relation to Rickett's Esthetic line will be measured in millimeter (mm).
Stability of dentition | 1 year post debond of orthodontic fixed appliances
  Any irregularity at lower labial segment will be measured using Little Irregularity Index. This will be measured in millimeter (mm).
Changes in arches parameters | 1 year post debond of orthodontic fixed appliances
  Intra arch changes will be measure based on intermolar width, intercanine width, arch length, overbite and overjet. This will be measured in millimeter (mm).
Impact of retainers on Oral Health Related Quality of Life | 1 year post debond of orthodontic fixed appliances
  Patients perception towards retainer will be measured using an Oral Health Related Quality of Life (OHIP) questionnaire. Patients will be assessed on how often they experienced the problems mentioned in the questionnaire throughout the time they use the retainers. The scale will be recorded as very often, quite often, sometimes, never, don't know.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Norhidayah@Nor Zahidah Mohd Tahir, MOrth, Principal Investigator — Faculty of Dentistry University of Malaya Kuala Lumpur
Locations (1):
- Faculty of Dentistry University of Malaya, Petaling Jaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lew K. Profile changes following orthodontic treatment of bimaxillary protrusion in adults with the Begg appliance. Eur J Orthod. 1989 Nov;11(4):375-81. doi: 10.1093/oxfordjournals.ejo.a036009. PMID 2591485
- [Result] Ab Rahman N, Low TF, Idris NS. A survey on retention practice among orthodontists in Malaysia. Korean J Orthod. 2016 Jan;46(1):36-41. doi: 10.4041/kjod.2016.46.1.36. Epub 2016 Jan 25. PMID 26877981
- [Result] Keating PJ. The treatment of bimaxillary protrusion. A cephalometric consideration of changes in the inter-incisal angle and soft tissue profile. Br J Orthod. 1986 Oct;13(4):209-20. PMID 3465369
- [Result] Shawesh M, Bhatti B, Usmani T, Mandall N. Hawley retainers full- or part-time? A randomized clinical trial. Eur J Orthod. 2010 Apr;32(2):165-70. doi: 10.1093/ejo/cjp082. Epub 2009 Oct 1. PMID 19797411
- [Result] Thickett E, Power S. A randomized clinical trial of thermoplastic retainer wear. Eur J Orthod. 2010 Feb;32(1):1-5. doi: 10.1093/ejo/cjp061. Epub 2009 Oct 14. PMID 19828592
- [Result] Gill DS, Naini FB, Jones A, Tredwin CJ. Part-time versus full-time retainer wear following fixed appliance therapy: a randomized prospective controlled trial. World J Orthod. 2007 Fall;8(3):300-6. PMID 17902334
- [Derived] Maskim N, Mohd Tahir NNZ, Wan Hassan WN. A randomized controlled trial comparing retainers in bimaxillary proclination cases. Clin Oral Investig. 2025 Feb 6;29(2):117. doi: 10.1007/s00784-025-06199-3. PMID 39912971